CLINICAL TRIAL: NCT01222637
Title: Dose-escalation, PK- and Safety Study With Single Agent CetuGEX™ in Patients With EGFR Positive Locally Advanced and/or Metastatic Cancer
Brief Title: CetuGEX™: Phase 1 Study in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEXMab52101
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumors
Keywords: advanced solid cancers; metastatic solid cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CetuGEX™, weekly (Experimental): application weekly
  Interventions: Drug: CetuGEX™
- CetuGEX™ 2-weekly (Experimental): application biweekly
  Interventions: Drug: CetuGEX™

INTERVENTIONS:
Drug: CetuGEX™
  Other Names: tomuzotuximab

SUMMARY:
This was a prospective, open label, multicenter study evaluating the safety, tolerability and pharmacokinetics of CetuGEX™ after intravenous administration in patients with EGFR positive, locally advanced and/or metastatic solid cancers. The effect of CetuGEX™ on the development of anti-drug antibodies and on tumour response was also evaluated.

DETAILED DESCRIPTION:
Male or female patients ≥18 years of age with a histologically confirmed locally advanced and/or metastatic solid organ tumor. Patients enrolled in Germany were required to have a positive EGFR overexpression status. Patients must have experienced a failure or non-availability of standard therapy (had received at least one line of chemotherapy and further standard therapy was not an option at study entry). Open-label, non-randomized, inter-patient dose-escalation, multi-center study. Patients were to receive CetuGEX until disease progression or until intolerable toxicities occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and age ≥ 18 yrs
2. Histologically confirmed EGFR positive locally advanced and/or metastatic solid organ tumour
3. Measurable or non-measurable tumour
4. Failure of standard therapy or non-availability of standard therapy (Patients must have received at least 1 line of chemotherapy and further standard therapy is not an option at study entry)
5. All anti-tumour therapies must be completed 4 weeks before start of study treatment; treatment with Cetuximab must be completed at least 6 weeks prior to study start
6. ECOG Performance Status ≤1 and estimated life expectancy of ≥ 3 months
7. Adequate organ function:

   * Bone marrow function: hemoglobin ≥ 100 g/L; white blood cell count (WBC) ≥ 3.0 x 10^9/L; absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; platelet count ≥ 100 x 10^9/L
   * Hepatic: aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤ 2.5 times upper limit of normal (ULN) (≤ 5 x ULN if hepatic metastases present); bilirubin ≤ 1.5 x ULN; alkaline phosphatase ≤ 5.0 x upper limit of normal (ULN)
   * Renal: creatinine < 1.5 x ULN
8. Patients of both genders with procreative potential must use effective contraception while enrolled in the study and for at least 4 weeks after the last study drug infusion
9. Written informed consent must be obtained prior to conducting any study-specific procedures

   For Expansion Phase only:
10. No prior treatment with Cetuximab allowed

Exclusion Criteria:

1. Chemotherapy, radiation, other anti-cancer therapies including any investigational agents at the study enrolment within 4 weeks prior to study enrolment
2. Concurrent anti-tumour therapy or concurrent immunotherapy
3. Concurrent systemic steroids except topical (inhaled, topical, nasal) or replacement therapy for the last 28 days.
4. Major surgery within 4 weeks prior entering the study and/or incomplete recovery from surgery or planned major surgery
5. Primary or secondary immune deficiency
6. Clinically active infections > CTCAE grade 2
7. Prior allergic reaction to a monoclonal antibody (e.g. Trastuzumab, Cetuximab or Bevacizumab).
8. Active hepatitis B assessed by serology, hepatitis C by histology; human immunodeficiency virus (HIV) seropositivity
9. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for ≥ 3 years will be allowed to enter the study.
10. Uncontrolled medical condition considered as high risk for the treatment with an investigational drug including unstable diabetes mellitus, vena-cava-syndrome, chronic symptomatic respiratory disease.
11. Clinical signs of brain metastasis or leptomeningeal involvement
12. Symptomatic congestive heart failure (New York Heart Association [NYHA] 3 or 4); unstable angina pectoris within 6 months prior to enrollment; significant cardiac arrhythmia, or history of stroke or transient ischemic attack within 1 year.
13. Active drug abuse or chronic alcoholism
14. Pregnancy or Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAE) assessed with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0 | throughout the study until 28±2 days after last infusion
  TEAE were coded by use of Medical Dictionary for Regulatory Activities (MedDRA) version 13.1
Incidence of clinically relevant abnormal clinical laboratory parameters | from first infusion until 28±2 days following the last infusion
  graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0
Dose-limiting toxicities (DLT) | from first infusion until 28±2 days following the last infusion
  DLTs were defined as drug-related:
  * Hematological or non-hematological toxicity grade 3 (excl. rash) or 4 excluding inadequately treated nausea and vomiting;
  * In case of skin reaction (rash) grade 4
Changes of corrected QT interval (QTc) duration | from first infusion until 28±2 days following the last infusion
  by use of 12-lead electrocardiograms (ECG)
To define the recommended phase II dose and regimen | from first infusion until 28±2 days following the last infusion
  Defining a recommended dose for a Phase II study was possible based on the available PK data in combination with the safety and activity data for CetuGEX™

SECONDARY OUTCOMES:
Anti-Tumor Activity: Confirmed Best Overall Response Rates | From date of randomization until the date of first documented progression, assessed up to 60 months
  Assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. Tumors were measured by computed tomography (CT) scan or magnetic resonance imaging (MRI)
Anti-Tumor Activity: Clinical Benefit Rates | From date of randomization until the date of first documented progression, assessed up to 60 months
  Assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. Tumors were measured by computed tomography (CT) scan or magnetic resonance imaging (MRI)
Eastern Cooperative Oncology Group (ECOG) Performance Status | From date of randomization until 28 days ± 2 days after the end of treatment
  The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The scale comprises six grades:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
Pharmacokinetics (PK): Area under the serum concentration-time curve (AUC) | Prior to 1st infusion, end of 1st infusion, 4 hours after end, 72 and 168 hours after start of 1st infusion, then before and after each infusion up to 10 weeks
  PK of CetuGEX™ after single and multiple administration
Pharmacokinetics (PK): Maximum serum concentration (Cmax) | Prior to 1st infusion, end of 1st infusion, 4 hours after end, 72 and 168 hours after start of 1st infusion, then before and after each infusion up to 10 weeks
  PK of CetuGEX™ after single and multiple administration
Pharmacokinetics (PK): Time to maximum serum concentration (tmax) | Prior to 1st infusion, end of 1st infusion, 4 hours after end, 72 and 168 hours after start of 1st infusion, then before and after each infusion up to 10 weeks
  PK of CetuGEX™ after single and multiple administration
Pharmacokinetics (PK): Minimal serum concentration (Cmin) | Prior to 1st infusion, end of 1st infusion, 4 hours after end, 72 and 168 hours after start of 1st infusion, then before and after each infusion up to 10 weeks
  PK of CetuGEX™ after single and multiple administration
Pharmacokinetics (PK): Terminal elimination half-life (t1/2) | Prior to 1st infusion, end of 1st infusion, 4 hours after end, 72 and 168 hours after start of 1st infusion, then before and after each infusion up to 10 weeks
  PK of CetuGEX™ after single and multiple administration
Pharmacokinetics (PK): Clearance rate (CL) | Prior to 1st infusion, end of 1st infusion, 4 hours after end, 72 and 168 hours after start of 1st infusion, then before and after each infusion up to 10 weeks
  PK of CetuGEX™ after single and multiple administration
Pharmacokinetics (PK): Volume of distribution (Vz) | Prior to 1st infusion, end of 1st infusion, 4 hours after end, 72 and 168 hours after start of 1st infusion, then before and after each infusion up to 10 weeks
  PK of CetuGEX™ after single and multiple administration

CONTACTS AND LOCATIONS:
Overall Officials: Glycotope GmbH, Study Director — Glycotope GmbH
Locations (4):
- Germany (2):
  - Glycotope Investigational Site, Hamburg
  - Glycotope Investigational Site, Heidelberg
- Glycotope Investigational Site, Milan, Italy
- Glycotope Investigational Site, Bellinzona, Switzerland

REFERENCES:
- [Result] Fiedler W, Cresta S, Schulze-Bergkamen H, De Dosso S, Weidmann J, Tessari A, Baumeister H, Danielczyk A, Dietrich B, Goletz S, Zurlo A, Salzberg M, Sessa C, Gianni L. Phase I study of tomuzotuximab, a glycoengineered therapeutic antibody against the epidermal growth factor receptor, in patients with advanced carcinomas. ESMO Open. 2018 Feb 1;3(2):e000303. doi: 10.1136/esmoopen-2017-000303. eCollection 2018. PMID 29464112